CLINICAL TRIAL: NCT03764150
Title: Factors Associated With Hypoventilation in the Myotonic Dystrophy, Progressive Profile Over 5 Years
Acronym: Steinert
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_04/0923; 2009-A00588-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-11-19; First posted 2018-12-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Myotonic Dystrophy, Steinert
Keywords: Sleep Apnea Syndrome; Muscular Diseases; non invasive ventilation; Diaphragmatic Disorder
MeSH Terms: conditions — Myotonic Dystrophy; Sleep Apnea Syndromes; Muscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PaCO2> 45 mmHg: Diurnal hypercapnia defined by PaCO2> 45 mmHg
- PaCO2 <45 mmHg: PaCO2 diurnal within the limits of normal (PaCO2 <45 mmHg)

SUMMARY:
The aim of this study is to determine the factors associated with alveolar hypoventilation in terms of cognitive impairment, daytime sleepiness, respiratory function, nocturnal respiratory events This evaluation will clarify the clinical phenotypes of respiratory disease in myotonic steinert dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Myotonic dystrophy of Steinert genetically confirmed (number of known CTG repeats), in its classical form of adult

Exclusion Criteria:

* Inability to perform EFR assessment or polysomnography
* Moderate to severe asthma according to the GINA classification
* moderate to severe COPD (> stage 1 of the GOLD recommendations)
* Other significant respiratory pathology
* Patient already on NIV, CPAP or under oxygen therapy
* Impossibility of receiving enlightened information
* Inability to participate in the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with a myotonic dystrophy of Steinert who consults in pneumology and who will have Respiratory functional exploration
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2010-06-30 (Actual); Primary Completion 2023-06-11 (Actual); Study Completion 2023-06-11 (Actual)

PRIMARY OUTCOMES:
Change of measurement of spirometry | every year during 5 years
  composite predictive factors of alveolar hypoventilation
Change respiratory force | every year during 5 years
  composite predictive factors of alveolar hypoventilation to change Inspiratory and expiratory force
Change CO2 response (Read test) | every year during 5 years
  composite predictive factors of alveolar hypoventilation
Change subjective sleepiness (Epworth) | every year during 5 years
  composite predictive factors of alveolar hypoventilation
change Krupp's Fatigue Severity Scale (KFSS) | every year during 5 years
  composite predictive factors of alveolar hypoventilation This is a short questionnaire of 9 questions to which the patient responds on a Likert scale ranging from 1 to 7
change cognitive impairment by Trail Making Test A & B | every year during 5 years
  composite predictive factors of alveolar hypoventilation Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.
change Oximetry | every year during 5 years
  composite predictive factors of alveolar hypoventilation

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Perez, MD, Principal Investigator — University Hospital, Lille
Locations (6):
- France (6):
  - Centre Hospitalier Regional D' Angers, Angers
  - Ap-Hp Hu Paris Site Raymond Poincare, Garches
  - Hôpital Calmette, CHRU, Lille
  - Chu Montpellier, Montpellier
  - Chu de Nantes :Site Hôtel-Dieu- Hme - Nantes 1, Nantes
  - Ap-Hp Hu Pitie Salpetriere, Paris

IPD SHARING:
Plan to Share IPD: No